CLINICAL TRIAL: NCT03075462
Title: An Open, Non-randomised, Multi-centre Phase I Study to Assess the Safety and Efficacy of Fluzoparib Given in Combination With Apatinib in Patients With Recurrent Ovarian Cancer or Triple Negative Breast Cancer
Brief Title: A Study of Fluzoparib Given in Combination With Apatinib in Ovarian or Breast Cancer Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Collaborators: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FZPL-I-104-OC/BC
Record Dates: First submitted 2017-03-06; First posted 2017-03-09 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Ovarian Cancer; Triple Negative Breast Cancer
Keywords: PARP inhibitor; VEGFR inhibitor; Combination therapy; Ovarian Cancer; Triple Negative Breast Cancer
MeSH Terms: conditions — Ovarian Neoplasms; Triple Negative Breast Neoplasms | interventions — fluzoparib; apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fluzoparib + Apatinib (Experimental): Fluzoparib and apatinib will be separately administered to patients on the 1st and 4th day, respectively. Then from the 7th day they are administered continuously and orally in combination, 28 days per cycle, until disease progression or unacceptable toxicity.
  Interventions: Drug: Fluzoparib; Drug: Apatinib

INTERVENTIONS:
Drug: Fluzoparib — Fluzoparib either at 40,60,80mg twice daily,capsule oral.
  Other Names: SHR3162; HS10160
Drug: Apatinib — Apatinib at 250mg once daily, tablet oral

SUMMARY:
Fluzoparib is an oral potent, selective poly-ADP ribose polymerase-1 (PARP-1) and PARP-2 inhibitor; Apatinib is an oral selective vascular endothelial growth factor receptor (VEGFR) inhibitor. This open-label, dose finding phase I trial studies the tolerability and the best dose of fluzoparib in combination with apatinib and to see how well these two drugs work together in the treatment of patients with recurrent ovarian cancer or triple negative breast cancer. The safety and efficacy of fluzoparib in combination with apatinib will be explored. Both dose escalation and dose expansion parts are included in this study.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
* Life expectancy of more than 12 weeks.
* Histologically or cytologically confirmed high-grade papillary-serous epithelial ovarian cancer，primary peritoneal, or fallopian tube cancers; subjects with a known deleterious breast cancer gene (BRCA) mutation and any other high-grade histology are also eligible. Subjects should have platinum-sensitive disease, where platinum-sensitive disease is defined as having had a > 6 month interval since last receiving platinum therapy prior to disease recurrence. Additionally, subjects with histologically or cytologically confirmed triple negative breast cancer (TNBC）, that is locally advanced or metastatic, are also eligible.
* Prior therapy：subjects with ovarian cancer，primary peritoneal, or fallopian tube cancers have received only 2 lines of platinum-based chemotherapies, and TNBC patients have received only 1 line of standard chemotherapy. Each prior chemotherapy must be given for at least 2 cycles.
* At least one measurable lesion that can be accurately assessed by imaging (CT/MRI) at baseline
* Subjects who have overall good overall general condition.
* Signed informed consent.

Exclusion Criteria:

* Subjects who received any previous treatment with any PARP inhibitors.
* Subjects who received any previous treatment with any VEGFR inhibitors.
* Less than 4 weeks from the last clinical trial.
* Less than 4 weeks from the last radiotherapy, chemotherapy, surgery, hormone treatment and target therapy.
* Unstable or uncontrolled hypertension.
* Subjects that are unable to swallow, or dysfunction of gastrointestinal absorption.
* Subjects with brain metastases.
* Subjects with uncontrolled hypokalemia and hypomagnesemia before study entry.
* Subjects with a known hypersensitivity to fluzoparib, apatinib or any of the excipients of the products.
* Ongoing infection (determined by investigator).
* History of immunodeficiency, including HIV-positive, suffering from other acquired, congenital immunodeficiency disease, or history of organ transplantation.
* Pregnant or breast-feeding women.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2017-03-09 (Actual); Primary Completion 2021-08-22 (Actual); Study Completion 2021-12-13 (Actual)

PRIMARY OUTCOMES:
The type and incidence of adverse events [safety and tolerability] | From screening up to 28 days after end of treatment
  Adverse events defined according to Common Terminology for Adverse Events (CTCAE) v4.03

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 24 months (approx) from the start of treatment
  [Complete response + Partial response (CR+PR)] based on RECIST 1.1
Disease Control Rate (DOR) | 24 months (approx) from the start of treatment
  [Complete response + Partial response + Stable disease (CR+PR+SD)] based on RECIST 1.1
Time to Progression (TTP) | From date of enrollment until the date of first objective progression or CA-125 progression (only for ovarian cancer patients), assessed up to 36 months
  The time from start of the treatment until radiographic disease progression or CA-125 progression specific for ovarian cancer patients
Overall Survival (OS) | From Cycle 1, Day 1 until death or up to 48 months (approx)
  Time from start of fluzoparib treatment until death due to any cause
Cmax | From the start of fluzoparib treatment alone to Cycle 2, Day 1 of combined treatment
  Maximum Plasma Concentration
T1/2 (Half-life) | From the start of fluzoparib treatment alone to Cycle 2, Day 1 of combined treatment
  The time required for the plasma concentration of a drug to be reduced by 50%
Area under curve (AUC) | Within the first 5 weeks from start of fluzoparib treatment
  Area under the plasma concentration-time curve
V/F | From the start of fluzoparib treatment alone to Cycle 2, Day 1 of combined treatment
  Volume of distribution
CL/F | From the start of fluzoparib treatment alone to Cycle 2, Day 1 of combined treatment
  Plasma Clearance

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hosptial, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Liu Y, Wang W, Yin R, Zhang Y, Zhang Y, Zhang K, Pan H, Wang K, Lou G, Li G, Zhang R, Li K, Rao J, Zhang B, Wang Y, Wang Q, Gao Y, Li H. A phase 1 trial of fuzuloparib in combination with apatinib for advanced ovarian and triple-negative breast cancer: efficacy, safety, pharmacokinetics and germline BRCA mutation analysis. BMC Med. 2023 Sep 29;21(1):376. doi: 10.1186/s12916-023-03046-8. PMID 37775744